CLINICAL TRIAL: NCT04904224
Title: Use of Pan-intestinal Capsule Endoscopy for Detection of Inflammatory Bowel Disease in the Case of Increased Fecal Calprotectin
Brief Title: Diagnosis of Inflammatory Bowel Disease by Examining the Entire Bowel by Pan-intestinal Capsule Endoscopy
Acronym: PEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Robert Bosch Medical Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Jorg G. Albert, Prof. Dr. med., Robert Bosch Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KKF-06-2019
Record Dates: First submitted 2021-05-22; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Inflammatory Bowel Diseases; Morbus Crohn
Keywords: Abdominal Pain; Diarrhea; Video Capsule Endoscopy; Panintestinal Video Capsule Endoscopy; Fecal Calprotectin
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Abdominal Pain; Diarrhea | interventions — Endoscopy; Colonoscopy

STUDY DESIGN:
Intervention Model Description: Randomized multicentric open-label study in cooperation with local gastroenterological specialist practices. A comparison is made of pan-intestinal capsule endoscopy versus colonoscopy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PICE (Active Comparator): Participants receive a panintestinal video capsule endoscopy (PICE)
  Interventions: Device: Panintestinal video capsule endoscopy
- Colonoscopy (Active Comparator): Participants receive an (Ileo-)Colonoscopy
  Interventions: Device: Colonoscopy

INTERVENTIONS:
Device: Panintestinal video capsule endoscopy — Performing a video capsule endoscopy using the Pill Cam Crohn's capsule from Medtronic
  Other Names: PillCam Crohn's Capsule
  Arms: PICE
Device: Colonoscopy — Performing a standard colonoscopy using the colonoscope available in the study center
  Other Names: (Ileo-)Colonoscopy
  Arms: Colonoscopy

SUMMARY:
The aim of this study is to discover inflammatory changes in the gastrointestinal tract in adult patients with suspicion of a chronic inflammatory bowel disease (IBD) by examining the entire bowel, including the small intestine, by using a video capsule. The study compares the video capsule endoscopy with colonoscopy with the question of inflammation and patient satisfaction with the respective examinations.

The study is aimed at participants who present to a gastroenterologist because of their complaints like persistent abdominal pain or diarrhea. An infectious genesis and celiac disease must be ruled out in advance.

In addition, the determination of the fecal calprotectin (fCal) is necessary for this study. Fecal calprotectin is a stool marker for the severity of an inflammation of the gastrointestinal tract, an increased fecal calprotectin can be an initial indication for the presence of a chronic inflammatory bowel disease.

As mentioned above, participants will be examined in one of two ways: either with an examination of the small and large intestines using video capsule endoscopy in one examination (i.e. ,panintestinal capsule endoscopy', PICE) or a colonoscopy is performed as the standard treatment. Which of the two methods is used will be decided by lot, electronically controlled.

Colon cleansing is necessary in preparation for both examinations. The advantage of being assigned to the video capsule group is, in addition to showing the entire intestine in one examination, that no sedation is necessary for this examination.

In addition to the examination, participants have to fill out a questionnaire with information about their state of affairs, their well-being and their experience with the examination. After a period of six month the participants will be contact by phone to inquire about their current state of health.

DETAILED DESCRIPTION:
People who contact a gastroenterologist because of persistent complaints like abdominal pain or diarrhea are suspicious having an inflammatory bowel disease and maybe meet the eligibility requirements for the study.

After checking the inclusion and exclusion criteria further necessary data (medical history, secondary diagnoses, previous examinations, etc.) as well as laboratory parameters (especially signs of inflammation and fecal calprotectin) are collected. After being informed about the study and potential risks, all patients giving written informed consent and who meet the eligibility requirements will be randomized in an open-label manner (participant and investigator) in a 1:1 ratio to video capsule endscopy intervention or colonoscopy. A follow-up by phone to evaluate the state of health is planned after six months.

The study center and established specialist practices are responsible for the study inclusion.

There will be no recruitment by advertising. Only participants who are introducing themselves due to complaints are offered study participation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Apply one of the following

  * Chronic abdominal pain for at least 4 weeks, min. 3/10 points on a visual pain scale
  * Persistent diarrhea, Stool frequency of at least 4 per day
  * doctor visit due to the mentioned complaints
* Exclusion of an infectious genesis or coeliac disease by serological testing or duodenal biopsy, if necessary
* Consent to study participation
* Fecal calprotectin > 50 µg/g

Exclusion Criteria:

* Pregnancy
* metastasized malignoma
* terminal renal insufficiency, renal insufficiency requiring dialysis
* swallowing disorder
* age < 18 years
* lack of consent
* infectious genesis of symptomps
* coeliac disease
* Relative contraindication:

  * evidence of strictures, strictures or fistulas in the gastrointestinal tract in imaging or in high suggestive symptoms, e.g. Ileus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-03-07 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Evidence of inflammatory Alterations in the Gastrointestinal Tract | through study completion, an average of 1 year
  Detection of inflammatory changes using vidoe capsule endoscopy or colonoscopy

SECONDARY OUTCOMES:
Number of Diagnosis of a Chronic Inflammatory Bowel Disease | through study completion, an average of 1 year
  Diagnosis of inflammatory bowel disease depending on the examination findings of video capsule endoscopy or colonoscopy
Number of Participants with Indication for a Therapy because of the Examination findings | through study completion, an average of 1 year
  Indication for a surgical or drug therapy

CONTACTS AND LOCATIONS:
Overall Officials: Joerg G. Albert, Study Director — Robert Bosch Medical Center
Locations (6):
- Germany (6):
  - Praxis Gersemann, Ditzingen, Baden-Wurttemberg
  - Praxis Escher, Leonberg, Baden-Wurttemberg
  - Gastroenterologische Schwerpunktpraxis, Stuttgart, Baden-Wurttemberg
  - Robert Bosch Medical Center, Stuttgart, Baden-Wurttemberg
  - Gastroenterologie am Pragsattel, Stuttgart, Baden-Wurttemberg
  - Ambulante Gastroenterologie, Stuttgart, Baden-Wurttemberg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albert JG, Martiny F, Krummenerl A, Stock K, Lesske J, Gobel CM, Lotterer E, Nietsch HH, Behrmann C, Fleig WE. Diagnosis of small bowel Crohn's disease: a prospective comparison of capsule endoscopy with magnetic resonance imaging and fluoroscopic enteroclysis. Gut. 2005 Dec;54(12):1721-7. doi: 10.1136/gut.2005.069427. Epub 2005 Jul 14. PMID 16020490
- [Background] Albert JG, Kotsch J, Kostler W, Behl S, Kaltz B, Bokemeyer B, Dollinger MM, Haerting J, Fleig WE. Course of Crohn's disease prior to establishment of the diagnosis. Z Gastroenterol. 2008 Feb;46(2):187-92. doi: 10.1055/s-2007-963524. PMID 18253897
- [Background] Carroccio A, Iacono G, Cottone M, Di Prima L, Cartabellotta F, Cavataio F, Scalici C, Montalto G, Di Fede G, Rini G, Notarbartolo A, Averna MR. Diagnostic accuracy of fecal calprotectin assay in distinguishing organic causes of chronic diarrhea from irritable bowel syndrome: a prospective study in adults and children. Clin Chem. 2003 Jun;49(6 Pt 1):861-7. doi: 10.1373/49.6.861. PMID 12765980
- [Background] Cotter J, Dias de Castro F, Moreira MJ, Rosa B. Tailoring Crohn's disease treatment: the impact of small bowel capsule endoscopy. J Crohns Colitis. 2014 Dec;8(12):1610-5. doi: 10.1016/j.crohns.2014.02.018. Epub 2014 Mar 14. PMID 24631311
- [Background] Dionisio PM, Gurudu SR, Leighton JA, Leontiadis GI, Fleischer DE, Hara AK, Heigh RI, Shiff AD, Sharma VK. Capsule endoscopy has a significantly higher diagnostic yield in patients with suspected and established small-bowel Crohn's disease: a meta-analysis. Am J Gastroenterol. 2010 Jun;105(6):1240-8; quiz 1249. doi: 10.1038/ajg.2009.713. Epub 2009 Dec 22. PMID 20029412
- [Background] Fleiss JL, Tytun A, Ury HK. A simple approximation for calculating sample sizes for comparing independent proportions. Biometrics. 1980 Jun;36(2):343-6. PMID 26625475
- [Background] Hale M, McAlindon ME. Capsule endoscopy as a panenteric diagnostic tool. Br J Surg. 2014 Feb;101(3):148-9. doi: 10.1002/bjs.9321. Epub 2013 Nov 19. No abstract available. PMID 24254382
- [Background] Hale MF, Drew K, McAlindon ME, Sidhu R. The diagnostic accuracy of faecal calprotectin and small bowel capsule endoscopy and their correlation in suspected isolated small bowel Crohn's disease. Eur J Gastroenterol Hepatol. 2016 Oct;28(10):1145-50. doi: 10.1097/MEG.0000000000000696. PMID 27384306
- [Background] Hale MF, Sidhu R, McAlindon ME. Capsule endoscopy: current practice and future directions. World J Gastroenterol. 2014 Jun 28;20(24):7752-9. doi: 10.3748/wjg.v20.i24.7752. PMID 24976712
- [Background] Jensen MD, Nathan T, Rafaelsen SR, Kjeldsen J. Diagnostic accuracy of capsule endoscopy for small bowel Crohn's disease is superior to that of MR enterography or CT enterography. Clin Gastroenterol Hepatol. 2011 Feb;9(2):124-9. doi: 10.1016/j.cgh.2010.10.019. Epub 2010 Nov 5. PMID 21056692
- [Background] Jensen MD, Kjeldsen J, Nathan T. Fecal calprotectin is equally sensitive in Crohn's disease affecting the small bowel and colon. Scand J Gastroenterol. 2011 Jun;46(6):694-700. doi: 10.3109/00365521.2011.560680. Epub 2011 Apr 1. PMID 21456899
- [Background] May A, Albert J, Keuchel M, Moog G, Hartmann D. [Capsule endoscopy for the diagnosis of small bowel diseases. An updated statement by the endoscopy section of DGVS]. Z Gastroenterol. 2010 Dec;48(12):1384-404. doi: 10.1055/s-0029-1245788. Epub 2010 Nov 24. No abstract available. German. PMID 21108180
- [Background] Pennazio M, Spada C, Eliakim R, Keuchel M, May A, Mulder CJ, Rondonotti E, Adler SN, Albert J, Baltes P, Barbaro F, Cellier C, Charton JP, Delvaux M, Despott EJ, Domagk D, Klein A, McAlindon M, Rosa B, Rowse G, Sanders DS, Saurin JC, Sidhu R, Dumonceau JM, Hassan C, Gralnek IM. Small-bowel capsule endoscopy and device-assisted enteroscopy for diagnosis and treatment of small-bowel disorders: European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2015 Apr;47(4):352-76. doi: 10.1055/s-0034-1391855. Epub 2015 Mar 31. PMID 25826168
- [Background] Petruzziello C, Calabrese E, Onali S, Zuzzi S, Condino G, Ascolani M, Zorzi F, Pallone F, Biancone L. Small bowel capsule endoscopy vs conventional techniques in patients with symptoms highly compatible with Crohn's disease. J Crohns Colitis. 2011 Apr;5(2):139-47. doi: 10.1016/j.crohns.2010.12.004. Epub 2011 Jan 14. PMID 21453883
- [Background] Smalley W, Falck-Ytter C, Carrasco-Labra A, Wani S, Lytvyn L, Falck-Ytter Y. AGA Clinical Practice Guidelines on the Laboratory Evaluation of Functional Diarrhea and Diarrhea-Predominant Irritable Bowel Syndrome in Adults (IBS-D). Gastroenterology. 2019 Sep;157(3):851-854. doi: 10.1053/j.gastro.2019.07.004. Epub 2019 Jul 11. No abstract available. PMID 31302098
- [Background] Spada C, Hassan C, Galmiche JP, Neuhaus H, Dumonceau JM, Adler S, Epstein O, Gay G, Pennazio M, Rex DK, Benamouzig R, de Franchis R, Delvaux M, Deviere J, Eliakim R, Fraser C, Hagenmuller F, Herrerias JM, Keuchel M, Macrae F, Munoz-Navas M, Ponchon T, Quintero E, Riccioni ME, Rondonotti E, Marmo R, Sung JJ, Tajiri H, Toth E, Triantafyllou K, Van Gossum A, Costamagna G; European Society of Gastrointestinal Endoscopy. Colon capsule endoscopy: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2012 May;44(5):527-36. doi: 10.1055/s-0031-1291717. Epub 2012 Mar 2. PMID 22389230
- [Background] Spada C, Hassan C, Munoz-Navas M, Neuhaus H, Deviere J, Fockens P, Coron E, Gay G, Toth E, Riccioni ME, Carretero C, Charton JP, Van Gossum A, Wientjes CA, Sacher-Huvelin S, Delvaux M, Nemeth A, Petruzziello L, de Frias CP, Mayershofer R, Amininejad L, Dekker E, Galmiche JP, Frederic M, Johansson GW, Cesaro P, Costamagna G. Second-generation colon capsule endoscopy compared with colonoscopy. Gastrointest Endosc. 2011 Sep;74(3):581-589.e1. doi: 10.1016/j.gie.2011.03.1125. Epub 2011 May 20. PMID 21601200
- [Background] Stange EF. Colitis ulcerosa - Morbus Crohn. UNI-MED SCIENCE, 5. Auflage, 2016
- [Background] Wehkamp J, Gotz M, Herrlinger K, Steurer W, Stange EF. Inflammatory Bowel Disease. Dtsch Arztebl Int. 2016 Feb 5;113(5):72-82. doi: 10.3238/arztebl.2016.0072. PMID 26900160